CLINICAL TRIAL: NCT04781790
Title: French National Registry of Bone Marrow Failures: Prospective and Retrospective Database Associated to a Collection of Biological Samples: RIME Project
Brief Title: French National Registry of Bone Marrow Failures
Acronym: RIME
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI17045J
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Bone Marrow Failure Syndrome
Keywords: aplastic anemia; Fanconi anemia; blackfan diamond anemia; telomeropathies; inherited aplastic anemia; acquired aplastic anemia; medullary hypoplasia
MeSH Terms: conditions — Bone Marrow Failure Disorders; Anemia, Aplastic; Fanconi Anemia; Anemia, Diamond-Blackfan

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Laboratory of hematology, Saint Louis hospital, Paris, France (blood, bone marrow, skin)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Bone marrow failure: Standard of care of patients with bone marrow failure
  Interventions: Other: Bone Marrow Failure

INTERVENTIONS:
Other: Bone Marrow Failure — without interventional intervention . biological collection in the routine care Standard of care of patients with bone marrow failure.

SUMMARY:
This is a unique clinical and biological database that collects standardized clinical information during the management of all patients with bone marrow failure syndromes (BMF) in France (multicenter registry), from diagnosis and throughout follow-up during the natural history of the disease, treated or not. In parallel, biological samples (blood and/or bone marrow and/or skin) are collected during clinical care and are biobanked in Saint-Louis Hospital (Hematology laboratory) in order to be used in translational research related to bone marrow failure diseases.

This registry has two main objectives:

* Public health care evaluation and improvement: to assess the medical and social needs inherent to the management of these rare diseases; to precisely assess the level of diagnosis and management of bone marrow failure syndromes in France; to evaluate the impact and guidance of the French reference center guidelines for diagnosis and treatment; to evaluate the real-life efficacy and tolerance of any given specific treatments; to analyze treatment's cost-effectiveness according to each situation.
* Research:

  * Epidemiology: to determine the incidence, prevalence, and distribution of different bone marrow failure syndromes at the national level;
  * Biology: to better understand the pathophysiology of BMF; to identify and to study complications within each entity, such as mechanisms underlying clonal evolution, new forms of inherited BMF and acute myeloid leukemia (AML)/MDS-predisposition syndromes, and to better and deeper characterize known entities;
  * Treatment: to identify prognostic factors and predictors of response; to identify side effects and impact of treatment on others organs and natural functions; to assess patients' quality of life as early as possible since diagnosis and throughout follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All age
* All diagnostic of BMF
* Having given his non-opposition to registry after understand overall aims
* Having signed a written informed consent (2 parents for patients aged less than 18) for collection of biological samples
* With health insurance coverage

Exclusion Criteria:

With myelodysplastic syndrome occurring in a patient over the age of 50 in absence of genetical predispositions, familial forms and history of medullary hypoplasia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with bone marrow failure syndromes (BMF)
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-02-06 (Actual); Primary Completion 2027-02-06 (Estimated); Study Completion 2027-02-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of bone marrow failure | at 10 years
Distribution of different bone marrow failure syndromes | at 10 years

SECONDARY OUTCOMES:
Quality of life assessed by EORTC QLQ-C30- v3 questionnaire | at inclusion
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
  EORTC QLQ-C30 Scoring Manual. Fayers PM et al. on behalf of the EORTC Quality of Life Group. EORTC, 2001. ISBN: 2-9300.
Quality of life assessed by EORTC QLQ-C30- v3 questionnaire | at 10 years
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
  EORTC QLQ-C30 Scoring Manual. Fayers PM et al. on behalf of the EORTC Quality of Life Group. EORTC, 2001. ISBN: 2-9300.
mechanisms underlying a clonal evolution or AML/MDS syndroms | at 10 years
Proportion of patients with new forms of constitutional aplasias | at 10 years
Proportion of patients with complications within each entity | at 10 years
Prognostic factor ans treatment response | at 10 years
Pathophysiology of bone marrow failures | at 10 years
Global response to treatment | at 10 years
Incidence and outcome of extra hematological complications including solid tumors, fertility | within 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hématologie Greffe, Paris, France